CLINICAL TRIAL: NCT03004027
Title: Enhancing Psychological Self-help With Implementation Intentions for Those With Visible Skin Difference and Fear of Negative Evaluation
Brief Title: Enhancing Psychological Self-help With Implementation Intentions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sheffield (Other)
Responsible Party: Principal Investigator, Jessica Lane, Trainee Clinical Psychologist, University of Sheffield
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 147400
Record Dates: First submitted 2016-12-17; First posted 2016-12-28 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Social Anxiety
Keywords: health behaviour change; implementation intention; if then plan; skin condition; visible difference; self help
MeSH Terms: conditions — Skin Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Enhanced (Experimental): self help leaflet enhanced with implementation intentions
  Interventions: Other: Self help leaflet
- Standard (Active Comparator): self help leaflet standard (without implementation intentions)
  Interventions: Other: Self help leaflet
- Waiting list control (No Intervention): Baseline measures administered only. self help intervention will be made available once the study has finished.

INTERVENTIONS:
Other: Self help leaflet — Self help leaflet entitled 'Building confidence in social situations: A guide for people living with a visible skin differences'
  Arms: Enhanced; Standard

SUMMARY:
Individuals with visible conditions often report experiencing lowered social confidence and encountering intrusive reactions from others, yet relatively few targeted psychosocial self help interventions are available.

The investigators will conduct a randomised controlled trial to compare the efficacy of an adapted form of an existing self-help intervention with an enhanced version of the same intervention that incorporates if-then planning instructions (or 'implementation intentions') and a control condition that will receive support as usual. Participants who self-identify as having a visible condition affecting the skin or hair, or scarring to the skin that negatively affects their social confidence will be allocated to one of three conditions: augmented self-help, standard self help or control. The interventions will be delivered online and participants will complete psychometric outcome measures at two time points, four weeks apart.

It is hypothesised that participants who receive the augmented self help intervention will have a statistically significant decrease in fear of negative evaluation in comparison to both the standard self-help and support as usual control groups.

DETAILED DESCRIPTION:
The proposed research will take the form of a randomised controlled trial conducted in accordance with CONSORT guidelines (http://www.consort-statement.org). Data will be collected online using Qualtrics. Participants will be required to answer all fields on Qualtrics, as a way of managing potential missing data.

Participants will be randomly allocated to one of three groups: (i) psychological self-help augmented with implementation intentions, (ii) standard psychological self-help or (iii) a no intervention waiting list control. Qualtrics will be used to randomly allocate participants to one of the three groups.

A sample size analysis has been conducted and calculated assuming two measures, three groups, an alpha of 0.05, a power of 0.8, and an effect size of 0.25; a total sample size of 120 participants would be needed (i.e. 40 per group). Allowing for an attrition rate of 20%, 144 participants would need to be recruited (i.e. 48 per group). Although participants will be randomised to condition, it is best practice for any differences at baseline to be controlled for in analyses and thus a between factors repeated measure analysis of variance (ANOVA) will be conducted.

ELIGIBILITY:
Inclusion Criteria:

* Participants self-identify as having a visible skin difference
* Participants will be aged 18 years or over
* Participants will be fluent in the English language

Exclusion Criteria:

Participants will be excluded if they are currently receiving psychotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 326 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Change in Brief Fear of Negative Evaluation-II at four weeks (Carleton, Collimore, & Asmundson, 2007) | At baseline and four weeks

SECONDARY OUTCOMES:
Change in Generalised Anxiety Disorder 7 at four weeks | At baseline and four weeks

OTHER OUTCOMES:
Change in Patient Health Questionnaire 9 at four weeks | At baseline and four weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jessica C Lane, Principal Investigator — University of Sheffield
Locations (1):
- University of Sheffield, Sheffield, South Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Possibility that data will be used in future research. Individual participant data includes age, gender, description of visible skin difference and scores on the Brief Fear of Negative Evaluation, General Anxiety Disorder 7, Patient Health Questionnaire 9 questionnaires. Data will be obtained with agreement from the primary investigator Jessica Lane (jlane1@sheffield.ac.uk)

REFERENCES:
- [Background] Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007 May;39(2):175-91. doi: 10.3758/bf03193146. PMID 17695343